CLINICAL TRIAL: NCT03673930
Title: The Acute and Chronic Cognitive and Cerebral Blood Flow Effects of Zanthozylum Armatum Fruit Extract: a Double Blind, Randomized, Placebo Controlled, Parallel Groups Study in Healthy Humans
Brief Title: Cognitive and Cerebral Blood Flow Effects of Zanthozylum Armatum Fruit Extract in Healthy Adults Aged 30 - 55
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Mibelle AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 53BS1
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Cognitive Change
Keywords: NIRS; mood; cognitive performance; Zanthozylum armatum; Nepalese pepper

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zanthozylum armatum (Active Comparator): fruit extract
  Interventions: Dietary Supplement: Zanthozylum armatum
- Placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Zanthozylum armatum — Zanthozylum armatum MCT oil extract
  Arms: Zanthozylum armatum
Dietary Supplement: Placebo — sunflower oil matched for appearance
  Arms: Placebo

SUMMARY:
Zanthozylum armatum (Z. armatum)-otherwise known as Nepalese pepper, or timut-is an perennial shrub found in India and across Southeast Asia. Preparations of the bark, fruit and seeds of Z. armatum have been extensively used in traditional Indian medicine. Preliminary data have indicated that preparations of Z. armatum may also be beneficial to cognitive function. The study aims to investigate the effects acute and chronic consumption of Z. armatum on cognitive function and cerebral blood flow.

DETAILED DESCRIPTION:
Zanthozylum armatum (Z. armatum) is an perennial shrub found in India and across Southeast Asia. Preparations of the bark, fruit and seeds of Z. armatum have been extensively used in traditional Indian medicine. For example, the fruits and seeds have been employed as an aromatic tonic in fever and dyspepsia and the essential oil of the fruits has exhibited antibacterial, antifungal and anthelmintic properties. Furthermore, the dried fruits are used as spice, especially in Nepalese and Sichuan cuisine with increasing popularity across Europe. With regard to physiological effects relevant to brain function, Z. armatum has also been traditionally used as a cardio-depressant; these vasodilatory properties have recently being linked to its antagonistic effect on calcium ion channel function as demonstrated in isolated rabbit aorta tissue. In addition, the observed anti-inflammatory and antioxidant effects of preparations of Z. armatum may serve to beneficially impact cognition with chronic administration.

Although direct effects of Z. armatum on brain function have yet to be assessed; Zanthozylum fruit comprises one constituent of the traditional Japanese herbal medicine Daikenchuto (DKT) where some data do exist. In a series of trials investigating the effects of DKT on learning and memory function in mice, it was established that the extract of Zanthozylum fruit contained in DKT alone that was associated with reductions in escape latency in the Morris Water Maze task. Interestingly, the authors also revealed that it was the amide hydroxy-ɑ-sanshool (HAS) isolated from the Zanthozylum fruit extract that was associated with these effects, speculating that the effect of HAS on escape latencies was due to a facilitation effect of HAS on acetylcholine release.

Given the evidence of potentially relevant mechanisms of action and initial evidence of cognitive effects of HAS in murine models, the aim of this study is to assess the acute and chronic effects of Z. armatum on cognitive function, mood, and cerebral blood flow in healthy adults aged 30 to 55 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must self-assess themselves as being in good health
* Aged 30 to 55 years at the time of giving consent
* Are proficient in English equivalent to IELTS band 6 or above

Exclusion Criteria:

* Have any pre-existing medical condition/illness which will impact taking part in the study NOTE: the explicit exceptions to this are controlled (medicated) hypertension, arthritis, asthma, hay fever, high cholesterol and reflux-related conditions. There may be other, unforeseen, exceptions and these will be considered on a case-by-case basis; i.e. participants may be allowed to progress to screening if they have a condition/illness which would not interact with the active treatments or impede performance
* Are currently taking prescription medications or dietary supplements including omega fatty acids / fish oils NOTE: the explicit exceptions to this are hormone replacement treatments for female participants where symptoms are stable, those medications used in the treatment of arthritis, high blood pressure, high cholesterol and reflux-related conditions; and those taken 'as needed' in the treatment of asthma and hay fever. As above, there may be other instances of medication use which, where no interaction with the active treatments is likely, participants may be able to progress to screening
* Have planned a surgery requiring general anaesthesia
* Have high blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg)
* Have a Body Mass Index (BMI) outside of the range 18-35 kg/m2
* Are pregnant, seeking to become pregnant or lactating
* Have learning difficulties, dyslexia
* Have a visual impairment that cannot be corrected with glasses or contact lenses (including colour-blindness)
* Smoker or regular consumption of nicotine containing products e.g. patches, gum, vaping
* Have a history of alcohol or drug abuse
* Excessive caffeine intake (>500 mg per day)
* Have food intolerances/sensitivities, especially against citrus fruits
* Have any health condition that would prevent fulfilment of the study requirements
* Are unable to complete all of the study assessments
* Are currently participating in other clinical or nutrition intervention studies, or have in the past 4 weeks
* Do not have a bank account (required for payment)
* Are non-compliant with regards treatment consumption

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Secondary memory score | Chronic (57 days)
  This is a composite measure derived from summing the z score performance on the following cognitive tasks: immediate word recall, delayed word recall, delayed picture recognition, delayed word recognition, delayed name to face recall (-1 to 1 where higher is better).

SECONDARY OUTCOMES:
STAI-trait total score | Baseline
  State-trait anxiety inventory 'trait' score (20-80; higher is more anxious)
STAI-state total score | Chronic (57 days)
  State-trait anxiety inventory 'state' score (20-80; higher is more anxious)
Secondary memory score | Acute (45, 180, 300 minutes post-dose)
  This is a composite measure derived from summing the z score performance on the following cognitive tasks: immediate word recall, delayed word recall, delayed picture recognition, delayed word recognition, delayed name to face recall (-1 to 1 where higher is better).
Secondary memory score | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  This is a composite measure derived from summing the z score performance on the following cognitive tasks: immediate word recall, delayed word recall, delayed picture recognition, delayed word recognition, delayed name to face recall (-1 to 1 where 1 is better).
Working memory score | Chronic (57 days)
  This is a composite measure derived from summing the z score performance on the numeric working memory task and Corsi block-tapping task (-1 to 1; where higher is better)
Working memory score | Acute (45, 180, 300 minutes post-dose)
  This is a composite measure derived from summing the z score performance on the numeric working memory task and Corsi block-tapping task (-1 to 1; where higher is better)
Working memory score | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  This is a composite measure derived from summing the z score performance on the numeric working memory task and Corsi block-tapping task (-1 to 1; where higher is better)
Speed of memory score | Acute (45, 180, 300 minutes post-dose)
  This is a composite measure derived from summing the z score reaction times on the numeric working memory task, the delayed name/face recall task, the delayed picture recognition task, and the delayed word recognition task (-1 to 1; where lower is better).
Speed of memory score | Chronic (57 days)
  This is a composite measure derived from summing the z score reaction times on the numeric working memory task, the delayed name/face recall task, the delayed picture recognition task, and the delayed word recognition task (-1 to 1; where lower is better)
Speed of memory score | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  This is a composite measure derived from summing the z score reaction times on the numeric working memory task, the delayed name/face recall task, the delayed picture recognition task, and the delayed word recognition task (-1 to 1; where lower is better).
Accuracy of attention score | Acute (45, 180, 300 minutes post-dose)
  This is a composite measure derived from summing the z score accuracy performance on the choice reaction time and Rapid visual information processing tasks (-1 to 1; where higher is better)
Accuracy of attention score | Chronic (57 days)
  This is a composite measure derived from summing the z score accuracy performance on the choice reaction time and Rapid visual information processing tasks (-1 to 1; where higher is better)
Accuracy of attention score | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  This is a composite measure derived from summing the z score accuracy performance on the choice reaction time and Rapid visual information processing tasks (-1 to 1; where higher is better)
Speed of attention score | Acute (45, 180, 300 minutes post-dose)
  This is a composite measure derived from summing the z score reaction times on the choice reaction time and Rapid visual information processing tasks (-1 to 1; where lower is better)
Speed of attention score | Chronic (57 days)
  This is a composite measure derived from summing the z score reaction times on the choice reaction time and Rapid visual information processing tasks (-1 to 1; where lower is better)
Speed of attention score | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  This is a composite measure derived from summing the z score reaction times on the choice reaction time and Rapid visual information processing tasks (-1 to 1; where lower is better)
Immediate word recall task correctly identified words | Acute (45, 180, 300 minutes post-dose)
  total number (0-15; where higher is better)
Immediate word recall task correctly identified words | Chronic (57 days)
  total number (0-15; where higher is better)
Immediate word recall task correctly identified words | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  total number (0-15; where higher is better)
Immediate word recall task error responses | Acute (45, 180, 300 minutes post-dose)
  total number (can be any number; lower is better)
Immediate word recall task error responses | Chronic (57 days)
  total number (can be any number; lower is better)
Immediate word recall task error responses | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  total number (can be any number; lower is better)
Delayed word recall task correctly identified words | Acute (45, 180, 300 minutes post-dose)
  total number (0-15; where higher is better)
Delayed word recall task correctly identified words | Chronic (57 days)
  total number (0-15; where higher is better)
Delayed word recall task correctly identified words | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  total number (0-15; where higher is better)
Delayed word recall task correctly error responses | Acute (45, 180, 300 minutes post-dose)
  total number (can be any number; lower is better)
Delayed word recall task correctly error responses | Chronic (57 days)
  total number (can be any number; lower is better)
Delayed word recall task correctly error responses | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  total number (can be any number; lower is better)
Picture recognition accuracy | Acute (45, 180, 300 minutes post-dose)
  (%; 0-100; where higher is better)
Picture recognition accuracy | Chronic (57 days)
  (%; 0-100; where higher is better)
Picture recognition accuracy | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  (%; 0-100; where higher is better)
Picture recognition reaction time | Acute (45, 180, 300 minutes post-dose)
  (ms; lower is better)
Picture recognition reaction time | Chronic (57 days)
  (ms; lower is better)
Picture recognition reaction time | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  (ms; lower is better)
Word recognition accuracy | Acute (45, 180, 300 minutes post-dose)
  (%; 0-100; where higher is better)
Word recognition accuracy | Chronic (57 days)
  (%; 0-100; where higher is better)
Word recognition accuracy | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  (%; 0-100; where higher is better)
Word recognition reaction time | Acute (45, 180, 300 minutes post-dose)
  (ms; lower is better)
Word recognition reaction time | Chronic (57 days)
  (ms; lower is better)
Word recognition reaction time | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  (ms; lower is better)
Name to face recall correct responses | Acute (45, 180, 300 minutes post-dose)
  number (0-24; higher is better)
Name to face recall correct responses | Chronic (57 days)
  number (0-24; higher is better)
Name to face recall correct responses | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  number (0-24; higher is better)
Name to face recall reaction time | Acute (45, 180, 300 minutes post-dose)
  (ms; lower is better)
Name to face recall reaction time | Chronic (57 days)
  (ms; lower is better)
Name to face recall reaction time | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  (ms; lower is better)
Peg and ball task planning time | Acute (45, 180, 300 minutes post-dose)
  (ms; lower is better)
Peg and ball task planning time | Chronic (57 days)
  (ms; lower is better)
Peg and ball task planning time | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  (ms; lower is better)
Peg and ball task completion time | Acute (45, 180, 300 minutes post-dose)
  (ms; lower is better)
Peg and ball task completion time | Chronic (57 days)
  (ms; lower is better)
Peg and ball task completion time | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  (ms; lower is better)
Peg and ball task errors | Acute (45, 180, 300 minutes post-dose)
  number (can be any number, lower is better)
Peg and ball task errors | Chronic (57 days)
  number (can be any number, lower is better)
Peg and ball task errors | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  number (can be any number, lower is better)
Corsi blocks accuracy | Acute (45, 180, 300 minutes post-dose)
  Average scores from the last five correctly completed trials from the corsi block-tapping task
Corsi blocks accuracy | Chronic (57 days)
  Average scores from the last five correctly completed trials from the corsi block-tapping task
Corsi blocks accuracy | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  Average scores from the last five correctly completed trials from the corsi block-tapping task
Choice reaction time accuracy | Acute (45, 180, 300 minutes post-dose)
  (%; 0-100; where higher is better)
Choice reaction time accuracy | Chronic (57 days)
  (%; 0-100; where higher is better)
Choice reaction time accuracy | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  (%; 0-100; where higher is better)
Choice reaction time reaction time | Acute (45, 180, 300 minutes post-dose)
  (ms; lower is better)
Choice reaction time reaction time | Chronic (57 days)
  (ms; lower is better)
Choice reaction time reaction time | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  (ms; lower is better)
Numeric working memory accuracy | Acute (45, 180, 300 minutes post-dose)
  (ms; lower is better)
Numeric working memory accuracy | Chronic (57 days)
  (%; 0-100; where higher is better)
Numeric working memory accuracy | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  (%; 0-100; where higher is better)
Numeric working memory reaction time | Acute (45, 180, 300 minutes post-dose)
  (ms; lower is better)
Numeric working memory reaction time | Chronic (57 days)
  (ms; lower is better)
Numeric working memory reaction time | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  (ms; lower is better)
Serial 3 subtractions total responses | Acute (45, 180, 300 minutes post-dose)
  number - calculated from the 3 cycles of the Cognitive Demand Battery; higher is better
Serial 3 subtractions total responses | Chronic (57 days)
  number - calculated from the 3 cycles of the Cognitive Demand Battery; higher is better
Serial 3 subtractions total responses | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  number - calculated from the 3 cycles of the Cognitive Demand Battery; higher is better
Serial 3 subtractions total error responses | Acute (45, 180, 300 minutes post-dose)
  number - calculated from the 3 cycles of the Cognitive Demand Battery; lower is better
Serial 3 subtractions total error responses | Chronic (57 days)
  number - calculated from the 3 cycles of the Cognitive Demand Battery; lower is better
Serial 3 subtractions total error responses | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  number - calculated from the 3 cycles of the Cognitive Demand Battery; lower is better
Serial 7 subtractions total responses | Acute (45, 180, 300 minutes post-dose)
  number - calculated from the 3 cycles of the Cognitive Demand Battery; higher is better
Serial 7 subtractions total responses | Chronic (57 days)
  number - calculated from the 3 cycles of the Cognitive Demand Battery; higher is better
Serial 7 subtractions total responses | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  number - calculated from the 3 cycles of the Cognitive Demand Battery; higher is better
Serial 7 subtractions total error responses | Acute (45, 180, 300 minutes post-dose)
  number - calculated from the 3 cycles of the Cognitive Demand Battery; lower is better
Serial 7 subtractions total error responses | Chronic (57 days)
  number - calculated from the 3 cycles of the Cognitive Demand Battery; lower is better
Serial 7 subtractions total error responses | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  number - calculated from the 3 cycles of the Cognitive Demand Battery; lower is better
Rapid visual information processing accuracy | Acute (45, 180, 300 minutes post-dose)
  (%) - calculated from the 3 cycles of the Cognitive Demand Battery (%; 0-100; where higher is better)
Rapid visual information processing accuracy | Chronic (57 days)
  (%) - calculated from the 3 cycles of the Cognitive Demand Battery (%; 0-100; where higher is better)
Rapid visual information processing accuracy | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  (%) - calculated from the 3 cycles of the Cognitive Demand Battery (%; 0-100; where higher is better)
Rapid visual information processing reaction time | Acute (45, 180, 300 minutes post-dose)
  (ms) - calculated from the 3 cycles of the Cognitive Demand Battery; lower is better
Rapid visual information processing reaction time | Chronic (57 days)
  (ms) - calculated from the 3 cycles of the Cognitive Demand Battery; lower is better
Rapid visual information processing reaction time | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  (ms) - calculated from the 3 cycles of the Cognitive Demand Battery; lower is better
Rapid visual information processing false alarms | Acute (45, 180, 300 minutes post-dose)
  number - calculated from the 3 cycles of the Cognitive Demand Battery; lower is better
Rapid visual information processing false alarms | Chronic (57 days)
  number - calculated from the 3 cycles of the Cognitive Demand Battery; lower is better
Rapid visual information processing false alarms | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  number - calculated from the 3 cycles of the Cognitive Demand Battery; lower is better
Mental fatigue | Acute (45, 180, 300 minutes post-dose)
  visual analogue scale (%) - calculated from the 3 cycles of the Cognitive Demand Battery (0-100; higher indicates more fatigue)
Mental fatigue | Chronic (57 days)
  visual analogue scale (%) - calculated from the 3 cycles of the Cognitive Demand Battery (0-100; higher indicates more fatigue)
Mental fatigue | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  visual analogue scale (%) - calculated from the 3 cycles of the Cognitive Demand Battery (0-100; higher indicates more fatigue)
Subjective mood - Alert | Acute (45, 180, 300 minutes post-dose)
  derived from Bond Lader visual analogue scales (0-100; higher is more alert)
Subjective mood - Alert | Chronic (57 days)
  derived from Bond Lader visual analogue scales (0-100; higher is more alert)
Subjective mood - Alert | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  derived from Bond Lader visual analogue scales (0-100; higher is more alert)
Subjective mood - Content (visual analogue scale) | Acute (45, 180, 300 minutes post-dose)
  derived from Bond Lader visual analogue scales (0-100 higher is more content)
Subjective mood - Content | Chronic (57 days)
  derived from Bond Lader visual analogue scales(0-100 higher is more content)
Subjective mood - Content | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  derived from Bond Lader visual analogue scales(0-100 higher is more content)
Subjective mood - Calm | Acute (45, 180, 300 minutes post-dose)
  derived from Bond Lader visual analogue scales (0-100 higher is more calm)
Subjective mood - Calm | Chronic (57 days)
  derived from Bond Lader visual analogue scale (0-100 higher is more calm)
Subjective mood - Calm (Bond Lader visual analogue scale) | Superimposed chronic (57 days plus 45, 180, 300 minutes post-dose)
  derived from Bond Lader visual analogue scale (0-100 higher is more calm)
Cerebral blood flow during performance of cognitive tasks | Acute (120, 150 minutes post-dose)
  Measured (in umol) using quantitative near infrared spectroscopy (higher indicates increased blood volume)
Cerebral blood flow during performance of cognitive tasks | Superimposed chronic (57 days plus 120, 150 minutes post-dose)
  Measured (in umol) using quantitative near infrared spectroscopy (higher indicates increased blood volume)
Cerebral blood flow at rest | Acute (120, 150 minutes post-dose)
  Measured (in umol) using quantitative near infrared spectroscopy (higher indicates increased blood volume)
Cerebral blood flow at rest | Chronic (57 days)
  Measured (in umol) using quantitative near infrared spectroscopy (higher indicates increased blood volume)
Cerebral blood flow at rest | Superimposed chronic (57 days plus 120, 150 minutes post-dose)
  Measured (in umol) using quantitative near infrared spectroscopy (higher indicates increased blood volume)

CONTACTS AND LOCATIONS:
Overall Officials: Philippa A Jackson, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria university, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilani SN, Khan AU, Gilani AH. Pharmacological basis for the medicinal use of Zanthoxylum armatum in gut, airways and cardiovascular disorders. Phytother Res. 2010 Apr;24(4):553-8. doi: 10.1002/ptr.2979. PMID 20041426
- [Background] Kalia NK, Singh B, Sood RP. A new amide from zanthoxylum armatum. J Nat Prod. 1999 Feb;62(2):311-2. doi: 10.1021/np980224j. PMID 10075770
- [Background] Nakamura T, Komai N, Isogami I, Ueno K, Ikegami F, Ono K, Yano S. Memory and learning-enhancing effect of Daikenchuto, a traditional Japanese herbal medicine, in mice.Journal of Natural Medicines 60(1): 64-67, 2006
- See also: Link to study site website — http://nutrition-neuroscience.co.uk